CLINICAL TRIAL: NCT01948141
Title: FGFR1 Amplification as A Predictor of Efficacy in A Biomarker-Driven Phase II Study of BIBF 1120 in Advanced Squamous Cell Lung Cancer Patients Who Have Failed Up to Two Prior Chemotherapeutic Regimens
Brief Title: Nintedanib in Treating Patients With Advanced Non-Small Cell Lung Cancer Who Have Failed Up to Two Previous Chemotherapy Regimens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 225512; NCI-2013-01618 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 225512 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Squamous Cell Lung Cancer; Stage III Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nintedanib) (Experimental): Patients receive nintedanib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: nintedanib

INTERVENTIONS:
Drug: nintedanib — Given PO
  Other Names: BIBF 1120; multitargeted tyrosine kinase inhibitor BIBF 1120; Tyrosine Kinase Inhibitor BIBF 1120; Vargatef

SUMMARY:
This phase II trial studies how well nintedanib works in treating patients with advanced non-small cell lung cancer who have failed up to two previous chemotherapy regimens. Nintedanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the 6-month progression-free survival (PFS) rate of fibroblast growth factor receptor 1 (FGFR1) amplified squamous cell lung cancer patients treated with BIBF 1120 (nintedanib).

SECONDARY OBJECTIVES:

I. Compare the 6-month PFS rate for the entire FGFR1 amplified group versus the FGFR1 non-amplified patients.

II. Compare the 6-month PFS rate for each FGFR1 amplified group (low, intermediate, and high) versus historical controls and FGFR1 non-amplified patients.

III. To assess the following endpoints overall and by FGFR1 group: PFS, overall survival (OS), confirmed tumor response rate, and adverse events.

TERTIARY OBJECTIVES:

I. The relation of FGFR1 gene copy number with PFS, OS, confirmed response rate, and adverse events.

II. The relationship fibroblast growth factor receptor (FGFR) polymorphisms with toxicity and efficacy.

OUTLINE:

Patients receive nintedanib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced histologically proven squamous cell carcinoma of the lung
* Patients who have failed at least 1 systemic chemotherapy regimen for metastatic disease, but not more than 2 regimens
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* The pathologic tissue is available to determine FGFR1 amplification status
* Presence of either evaluable disease or measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Absolute neutrophil count (ANC) >= 1500/uL
* Hemoglobin (HgB) >= 9 g/dL
* Platelets >= 100,000/uL
* Total bilirubin =< upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 1.5 x ULN (ALT and AST =< 2.5 x ULN is acceptable if there is liver metastasis)
* Calculated or measured creatinine clearance >= 45 mL/min
* Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment and have a negative serum or urine pregnancy test done =< 7 days prior to registration (for women of childbearing potential only)
* Life expectancy >= 12 weeks
* Willingness to provide the blood specimens as required by the protocol; please note that the willingness to participate pertains only to the patient and does not factor in the institution's ability to participate in any part of the translational component

Exclusion Criteria:

* Patients with any known endothelial growth factor receptor (EGFR) mutation and/or anaplastic lymphoma receptor tyrosine kinase (ALK) translocation
* Symptomatic, untreated, or uncontrolled central nervous system (CNS) metastases or seizure disorder; patients with asymptomatic CNS metastases treated with whole brain radiation (WBRT) or gamma knife radiosurgery (GKR) may be enrolled >= 1 week after completion of WBRT/GKR provided toxicities are =< Common Toxicity Criteria (CTC) grade I at the time of registration and/or controlled with dexamethasone 2 mg once daily for at least 5 days at the time of study treatment; patients with symptomatic CNS metastases treated with WBRT/GKR may be enrolled >= 2 weeks after completion of WBRT/GKR provided toxicities are =< CTC grade 1 at the time of registration and neurologic symptoms controlled with dexamethasone =< 2 mg once daily for at least 1 week at the time of study treatment
* Patients receiving palliative radiation to skeletal metastases may be registered as early as 1 week after completion of radiation therapy provided toxicities are =< CTC grade I at the time of registration
* Any of the following prior therapies for malignancy:

  * Systemic chemotherapy =< 4 weeks prior to registration
  * Radiation therapy =< 4 weeks prior to registration (exceptions noted in the prior bullet); the site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease
  * Major surgery (i.e., laparotomy), open biopsy, or significant traumatic injury =< 4 weeks prior to registration; minor surgery =< 2 weeks prior to registration; insertion of a vascular access device is not considered major or minor surgery in this regard
  * Other investigational agent =< 30 days prior to study treatment
* The following patients will be excluded from this study:

  * Pregnant women
  * Breastfeeding women
  * Men or women who are sexually active and unwilling to use a medically acceptable method of contraception (e.g., such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during the trial and for at least three months after end of active therapy; a highly effective method of birth control is defined as one which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly; patients will be considered to be of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation/salpingectomy, or post-menopausal for at least 2 years
* Second primary malignancy with the following exceptions which are allowed:

  * Carcinoma in situ of the cervix
  * Non-melanoma skin cancer
  * History of low-grade (Gleason score =< 6) localized prostate cancer even if diagnosed < 5 years prior to registration
  * Treated stage I breast cancer even if diagnosed =< 5 years prior to registration
  * Other prior malignancy (including melanoma) allowed if it was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of BIBF 1120 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or extensive small bowel resection)
* Leptomeningeal disease
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded because of possible pharmacokinetic interactions with oral investigational agents
* Unwilling to, or unable to, comply with the protocol
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring systemic antimicrobial therapy (including history of active or chronic hepatitis C and/or hepatitis B infection), significant pulmonary symptoms at baseline due to disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Centrally located tumors with radiographic evidence (computed tomography [CT] or magnetic resonance imaging [MRI]) of local invasion of major blood vessels
* Significant weight loss (> 10% of baseline body mass) within past 6 months prior to inclusion into the study
* Coagulation parameters: International normalized ratio (INR) > 2, prothrombin time (PT) and partial thromboplastin time (PTT) > 50% of deviation of institutional ULN
* Proteinuria by Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or greater
* Known inherited predisposition to bleeding or thrombosis
* Therapeutic anticoagulation (except for low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous device) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid < 325 mg per day)
* Baseline hemoptysis, per clinician/investigator evaluation
* Active alcohol or drug abuse
* History of arterial or venous thrombotic/embolic events =< 12 months prior to registration
* Prior history with BIBF 1120 or any other vascular endothelial growth factor (VEGF)/VEGF receptor (R) inhibitor
* New York Heart Association (NYHA) class III or IV; NOTE: patients classified as NYHA class II controlled with treatment may participate, with increased monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2016-08-16 (Actual); Study Completion 2016-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongbin Chen, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Nintedanib): Patients receive nintedanib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  nintedanib: Given PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Nintedanib)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression Free Survival (PFS) Rate Within the Entire FGFR1 Amplified Group
Description: The 6-month PFS rate was defined as the proportion of patients who were alive and progression-free at 6 months after start of study treatment. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: At 6 months
Population: All patients in FGFR1 amplified group
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 2
percentage of participants | 0 [0 to 65.8]

2. Secondary Outcome: Compare the 6-month PFS Rate for the Entire FGFR1 Amplified Group Versus the FGFR1 Non-amplified Patients.
Description: The 6-month PFS rate was defined as the proportion of patients who were alive and progression-free at 6 months after start of study treatment.
Time Frame: Time from study entry to the first of either disease progression or death, assessed at 6 months
Population: All treated and eligible patients. One participant was not done due to not enough tissue.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 5
percentage of participants
  Amplified | 0
  Non-amplified | 0
  Total | 0

3. Secondary Outcome: Compare the 6-month PFS Rate for Each FGFR1 Amplified Group (Low, Intermediate, and High) Versus FGFR1 Non-amplified Patients.
Description: as for outcome 2
Time Frame: Time from study entry to the first of either disease progression or death, assessed at 6 months
Population: All treated and eligible patients. One participant was not done due to not enough tissue.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 5
percentage of participants
  Non-amplified | 0
  Intermediate amplification | 0
  High amplificiation | 0
  Total | 0

4. Secondary Outcome: 6-month PFS Rate for Each of the FGFRI Amplified Groups (Low, Intermediate, High) in Comparison to Historical Controls
Description: as for outcome 2
Time Frame: Time from study entry to the first of either disease progression or death, assessed at 6 months
Population: No comparison was done do versus historical controls because it was inappropriate due to the small number of patients available.
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from study entry to death from any cause.
Time Frame: From study entry to death from any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 6
months
  Amplified | 10.2 [4 to 16.4]
  Non-amplified | 5.8 [4.6 to 23.7]
  Overall | 10.6 [4 to 23.7]
Statistical Analysis 1: Comparison: Treatment (Nintedanib); Test type: Superiority or Other; p = 0.59, Log Rank

6. Secondary Outcome: Tumor Response Rate
Description: Tumor Response rate was defined as the proportion of patients who had Complete Response (CR) or Partial Response (PR) by RECIST 1.1 Criteria. Complete Response (CR): Disappearance of all target lesions. Any lymph nodes must have a reduction in short axis to < 10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 3 years
Population: All treated and eligible patients. No statistics computed due to all patients were non-response in both groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 6
percentage of participants
  Amplified | 0 [0 to 66]
  Non-amplified | 0 [0 to 56]
  Total | 0 [0 to 39]

7. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: Percentage of participants with adverse events. Incidence of Adverse Events (AEs) was Accessed by the National Cancer Institute (NCI) CTCAE Version 4.0.
Time Frame: Up to 30 days post-treatment
Population: All treated and eligible patients. No statistics computed due to all patients had AEs in both groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 6
percentage of participants
  Total | 100 [61 to 100]
  Amplified | 100 [34 to 100]
  Non-amplified | 100 [44 to 100]

8. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) was defined as the time from study entry to the first of either disease progression or death.
Time Frame: Time from study entry to the first of either disease progression or death, assessed up to 3 years
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 6
months
  Overall | 2.7 [1.7 to 15.1]
  Amplified | 1.8 [1.8 to 1.9]
  Non-amplified | 3.4 [1.7 to 5.4]
Statistical Analysis 1: Comparison: Treatment (Nintedanib); Test type: Superiority or Other; p = 0.36, Log Rank

ADVERSE EVENTS:
Arm/Group | Treatment (Nintedanib)
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nintedanib) (N=6)
Septic shock (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nintedanib) (N=6)
Cardiac disorder (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (8)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 4 (5)
Pyrexia (General disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Blood alkaline phosphatase increased (Investigations) | 3 (5)
Gamma-glutamyltransferase increased (Investigations) | 2 (4)
Lymphocyte count increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes